CLINICAL TRIAL: NCT02610166
Title: Jointly Managing JIA Online: An Internet-based Psycho-educational Game for Children With Juvenile Idiopathic Arthritis (JIA) and Their Parents
Brief Title: Jointly Managing JIA Online: An Internet-based Psycho-educational Game for Children With JIA and Their Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Provincial Health Services Authority British Columbia (Other); Alberta Children's Hospital (Other); Montreal Children's Hospital of the MUHC (Other); IWK Health Centre (Other); Children's Hospital of Eastern Ontario (Other); St. Justine's Hospital (Other); University of Toronto (Other); McGill University (Other); University of Florida (Other); Children's Hospital of Western Ontario (Other); University of Kansas Medical Center (Other); Memorial University of Newfoundland (Other)
Responsible Party: Principal Investigator, Jennifer Stinson, Clinician Scientist/Clinical Nurse Specialist/NP, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000048447
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Game (Experimental): Access to the game.
  Interventions: Behavioral: Game
- Usual Care (Active Comparator): Control group.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Game — In addition to standard medical care, children in the experimental group will receive the Match-3 game. The game will be designed for short individual gameplay sessions (as little as a few seconds), once to three times a day, over the course of 8 weeks, involving no more than 15 minutes per day in anticipated screen time. There is no way to "lose" the game. Through a structured series of daily interactions, the player will learn strategies and develop decision-making abilities that will assist with management of their own JIA. The Match 3 concept (similar to the game, Bejeweled) will require the player to successfully match the treatment strategy to the JIA symptom.
  Arms: Game
Other: Usual Care — Children in usual care group receive standard medical care.
  Arms: Usual Care

SUMMARY:
Arthritis in children is a long-term illness and it can make a child's life very difficult. In children 8-11 years old, the child and their family work together to deal with the problems that arthritis can cause. Learning to cope with and manage the problems that come with arthritis can stop it from getting worse. It is important to create programs that teach children and families how to cope with and manage arthritis. This study will develop and test an online game that helps children learn how to better manage their arthritis. The goal of these studies is to test: (1) how easy to use and acceptable the online game is; and (2) if children who play the game feel less pain, have fewer limitations, and a better quality of life compared to children who do not play the game.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 8 and ≤ 11 years of age
2. Diagnosed with JIA (minimum 3 months) using International League of Associations for Rheumatology classification criteria96
3. Active disease
4. Child and primary parent/caregiver are able to speak and read English or French
5. Participants are willing and able to complete online measures

Exclusion Criteria:

1. Cognitive impairments (as assessed by reviewing medical chart and consultation with the patient's rheumatologist)
2. Major co-morbid illnesses (e.g., medical [inflammatory bowel disease, cancer, diabetes] or psychiatric [depression, anxiety]) which may impact their ability to understand and use the game or complete outcome assessments (as determined by their rheumatologist).
3. Children currently participating in other Cognitive Behavioural Therapy (CBT) interventions
4. Usability testing participants

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Participant Accrual | 8 weeks
  This will be centrally tracked by the clinical research project coordinator (CRPC).
Intervention Fidelity | 8 weeks
  Any issues or difficulties encountered during implementation of the intervention, control strategy, or outcome measures will be tracked throughout the study by the CRPC. For example, issues from a technical standpoint (for example, game not downloading properly, participant requiring assistance using the technology) or logistics standpoint.
Acceptability and Satisfaction with Intervention | 8 weeks
  Immediately post-trial children and parents in the intervention group will rate their acceptability of and satisfaction with the game and 10-15 English and 10-15 French children and one of their parents will take part in a brief qualitative interview.
Engagement with Intervention | 8 weeks
  Analytics will be used to track patterns of website program usage ("number of interactions" [clicks]).
Dropout Rates | 8 weeks
  This will be centrally tracked by the clinical research project coordinator (CRPC).

SECONDARY OUTCOMES:
Pain | 8 weeks
  Measured using the Standardized Universal Pain Evaluations for Rheumatology providers for children and youth (SUPERKIDZ). It consists of 4 domains: pain intensity and location (5 items), fatigue (1 item), pain interference/evaluative dimension (10 items), and affective/emotional dimension (4 items) for children ≥ 8 years (and parent proxy report for children 4-8 years). This measure takes 3 - 5 minutes to complete.
Pain-related Activity Limitations | 8 weeks
  Measured using the Child Activity Limitations Interview (CALI-21). This is a 21-item self-report scale divided into (i) active (e.g. gym, sports) and (ii) routine (e.g., schoolwork, reading) activity subscales.
Health-related Quality of Life | 8 weeks
  Measured using the Arthritis Pediatric Quality of Life Inventory (PedsQL). The PedsQL Arthritis Module is a 22-item self-report scale with five subscales: pain and hurt, daily activities, treatment, worry, and communication.
Self Efficacy | 8 weeks
  Measured using the Children's Arthritis Self-Efficacy Scale (CASE). The CASE is a disease specific 11-item self-report measure that is divided into three sub-scales: activity, symptom, and emotion. A 5-point Likert scale is used to rate responses to each item with 1 = "not at all sure" to 5 = "very sure" based on how confident the child is that they can manage disease effects.
JIA-specific Disease Knowledge | 8 weeks
  Measured using the 24-item Medical Issues, Exercise, Pain and Social Support Questionnaire (MEPS). MEPS is made up of 4 sub scales (medical issues, exercise, pain, and social support). Items are rated on a 10-cm VAS with higher scores indicating greater disease knowledge.
Adherence | 8 weeks
  Adherence to medical treatment will be assessed using the 34-item Child Adherence Report Questionnaire (CARQ) that assesses adherence to prescribed medications, exercises, and wearing of splints over the past 3 months. The CARQ was developed specifically for children with JIA and consists of three sections: (1) responsibility for treatment, (2) child's ability to adhere to the three types of treatment, and (3) perceptions about helpfulness of therapies. Items in the last two sections are rated on 11-point numeric pain rating scale with higher scores indicating better adherence and perceived helpfulness of therapies.

CONTACTS AND LOCATIONS:
Locations (7):
- Canada (7):
  - BC Children's Hospital, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec